CLINICAL TRIAL: NCT02154386
Title: Effect of Healing Time on New Bone Formation Following Tooth Extraction and Ridge Preservation With Demineralized Freeze-Dried Bone Allograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Brian L Mealey, Graduate Program Director, Periodontics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20130440H
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Bone Augmentation
Keywords: bone augmentation; tooth extraction; dental implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8-10 week healing group (Experimental): dental implant placed (and bone core biopsy harvested) 8-10 weeks after tooth extraction/grafting
  Interventions: Device: Ridge preservation using DFDBA
- 18-20 week healing group (Active Comparator): dental implant placed (and bone core biopsy harvested) 18-20 weeks after tooth extraction/grafting
  Interventions: Device: Ridge preservation using DFDBA

INTERVENTIONS:
Device: Ridge preservation using DFDBA — tooth extraction followed by ridge preservation grafting using DFDBA

SUMMARY:
Bone grafting following tooth extraction is commonly performed to preserve bony ridge dimensions adequate to support subsequent implant placement. Alveolar ridge resorption commonly occurs following tooth extraction, and the decrease in bone volume has the potential to make dental implant therapy impossible without surgery to reconstruct the ridge. The aim of ridge preservation grafting is to prevent or minimize this resorptive process, thereby preserving an adequate volume of bone for implant placement. Ridge preservation generally involves placement of a particulate bone graft material in the tooth socket, followed by use of a membrane or similar substance over the socket entrance to contain the bone graft. Various grafting materials have been recommended for these ridge preservation procedures, including demineralized freeze-dried bone allograft (DFDBA). The timing of dental implant placement following ridge preservation procedures is controversial, and few studies have examined the effects of different healing time intervals between ridge preservation and implant placement. The purpose of this project is to evaluate the formation of new bone at a site where tooth extraction has been performed followed by grafting using DFDBA. Two different study groups are included, one having the dental implant placed 8-10 weeks after tooth extraction and ridge grafting, the other having the dental implant placed 18-20 weeks after extraction and grafting.

DETAILED DESCRIPTION:
The purpose of this study is to compare healing following tooth extraction and ridge preservation with DFDBA at a healing time point 8-10 weeks after treatment compared to a healing time point 18-20 weeks after treatment. There have been no studies to determine differences in new bone formation using DFDBA for this purpose at various healing time points post-grafting. The primary objective is to histologically determine the amount of new bone formation and residual graft material present at the two healing time points after grafting with DFDBA. Histologic healing will be compared based on three criteria: % of new vital bone formation, % of residual graft material, and % of nonmineralized connective tissue/bone marrow. The null hypothesis is that there will be no difference between the % new bone formation at 8-10 weeks after grafting compared to 18-20 weeks after grafting.

This entire protocol involves procedures that are standard care. There will be two subject groups in this study. All subjects will require extraction of a non-molar tooth, followed by replacement of the missing tooth with a dental implant. In order to ensure that the bone core removed during implant osteotomy preparation is taken totally within the confines of the former tooth socket, the tooth to be extracted will have a position and angulation that is the same as the implant that will replace the tooth. Each group will have 22 subjects. Only one tooth will be evaluated in any given subject.

Both groups will consist of subjects who will have cortical DFDBA grafted into the extraction socket for ridge preservation following tooth extraction. Group 1 will have a biopsy core taken at the time of implant placement 8-10 weeks after socket grafting. Group 2 will have a biopsy core taken at the time of implant placement 18-20 weeks after socket grafting. Allocation of subjects into group 1 or 2 will based on randomization once enrolled into the study. Subjects will be asked to draw a sealed envelope out of a stack of envelopes, each containing a single slip of paper coded with #1 or a #2. This will determine the treatment group.

All of the bone graft materials used in this study will come from the same donor (LifeNet Health). The materials will be procured and processed in the same manner and will have the same particle size and percent residual calcium. This greatly decreases potential variability inherent in bone taken from different donors or processed in different manners.

At the time of subject enrollment, the following standard care procedures will be performed: Impressions will be made for fabrication of diagnostic casts and radiographs will be taken of the tooth to be extracted. A clear measurement stent will be made on the cast for vertical and horizontal ridge dimensions.

Following local anesthesia, the tooth will be extracted, and the number of bony walls in each socket will be recorded, along with the presence of any bony dehiscences or fenestrations. After extraction, the measurement stent will be placed and a hole will be made in the occlusal surface directly over the buccal bony wall and the lingual bony wall. Holes will be made in the buccal and lingual flanges of the measurement stent at a level approximately 3mm from the bony crests and ridge calipers will be used to make a horizontal ridge width measurement. These measurements will be recorded. The socket will be thoroughly debrided, a 1.0cc bottle of cortical DFDBA will be hydrated with sterile saline and the DFDBA will be placed in the socket to restore the ridge to appropriate contour. A collagen barrier (Collatape or Collaplug) will then be placed over the socket orifice and secured with sutures. Flaps will not be reflected to obtain primary closure. If a large dehiscence exists following extraction, which would most likely affect the facial socket wall, a collagen barrier with a longer resorption time, such as the Zimmer collagen socket repair membrane or BioGide collagen membrane will be used instead of Collatape or Collaplug. As part of standard care, patients will be prescribed systemic doxycycline 100mg twice a day for 7 days after surgery (if patient has sensitivity to doxycycline, alternate will be amoxicillin 500mg three times a day for 7 days). The patient will be seen 7-10 days after extraction/ridge preservation to assess healing, and again 1 month after the procedure.

The implant will be placed 8-10 weeks after ridge preservation in Group 1 and 18-20 weeks after ridge preservation in Group 2. At the time of implant placement, the first osteotomy will be prepared using a hollow trephine drill instead of a solid drill. Use of a hollow trephine allows retention of the bony core; whereas, use of solid drills results in removal of the bone in very small particles that cannot be examined histologically. Drilling of the pilot implant osteotomy has historically been done both ways (trephine drill or solid drill). The bone core in the trephine will be removed from the trephine, placed in 10% formalin, and prepared for histologic examination. The study will end immediately after removal of the trephined bone core.

Following initial preparation of the implant site with the trephine, the osteotomy will be completed and an implant of the appropriate length and diameter will be placed. The size of the implant will be such that it will engage not only newly formed bone in the socket itself, but at least 2-3mm of bone apical to the former socket site. A healing abutment will then be placed.

All subjects will be examined at 7-10 days and 1 month following implant placement. The patient will then be referred to their restorative dentist for final restoration.

The histologic cores will be processed for demineralized sections and will be stained. The following histologic parameters will be measured: percent new bone formation, percent residual graft material, and percent connective tissue/other.

ELIGIBILITY:
Inclusion Criteria:

* Patient currently a patient at dental school or eligible for treatment at dental school
* Patient resides within 50 mile radius of dental school
* A single rooted tooth that has been identified by dental faculty as requiring extraction
* Have adequate restorative space for a dental implant-retained restoration
* Have at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal.
* Have a dehiscence of the buccal or lingual bony plate of the tooth socket extending no more than 50% of the total depth of the socket.
* Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and non-pregnant women of child-bearing potential.

Exclusion Criteria:

* not meeting inclusion criteria above
* Active localized or systemic infection other than periodontitis.
* Inadequate bone dimensions or restorative space dimensions to place a dental implant
* Presence of a disease entity, medical condition or therapeutic regimen which decreases probability of soft tissue and bony healing, e.g., poorly controlled diabetes, chemotherapeutic and immunosuppressive agents, autoimmune diseases, history of bisphosphonate use or long-term steroid therapy.
* Positive medical history of endocarditis following oral or dental surgery.
* Sensitivity or allergy to Bacitracin, Gentamicin, Polymyxin B Sulfate, alcohol and/or surfactants (per package insert)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Health Science Center School of Dentistry, San Antonio, Texas, United States

REFERENCES:
- [Derived] Whetman J, Mealey BL. Effect of Healing Time on New Bone Formation After Tooth Extraction and Ridge Preservation With Demineralized Freeze-Dried Bone Allograft: A Randomized Controlled Clinical Trial. J Periodontol. 2016 Sep;87(9):1022-9. doi: 10.1902/jop.2016.160139. Epub 2016 Apr 30. PMID 27133791

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 8-10 Week Healing Group | 18-20 Week Healing Group
Started | 23 | 23
Completed | 22 | 21
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: The number of clinical measurements and core biopsies analyzed does not equal the number of subjects enrolled in each group because some subjects did not complete the study, some did not have core biopsy taken or biopsies were lost to processing issues, or some did not have clinical measurements taken at the time of implant placement
Groups:
- Total: Total of all reporting groups
Arm/Group | 8-10 Week Healing Group | 18-20 Week Healing Group | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Full Range); unit: years] | 56.1 [29 to 81] | 55.4 [23 to 81] | 55.7 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percent New Vital Bone Formation
Description: Bone core biopsy will be evaluated histologically for percent new vital bone formation
Time Frame: after removal of bone core from site of dental implant placement at 18-20 weeks following tooth extraction and grafting
Measure: Mean (Standard Deviation); unit: percentage of vital bone
Arm/Group | 8-10 Week Healing Group | 18-20 Week Healing Group
Number analyzed (Participants) | 20 | 19
percentage of vital bone | 32.63 (21.45) | 47.41 (11.66)

2. Secondary Outcome: Change in Ridge Width
Description: Ridge width measured at time of tooth extraction and grafting and again at time of implant placement. Changes in ridge width are determined (negative number signifies loss of ridge width)
Time Frame: at time of implant placement at 8-10 or 18-20 weeks following tooth extraction and grafting
Measure: Mean (Standard Deviation); unit: ridge width change (mm)
Arm/Group | 8-10 Week Healing Group | 18-20 Week Healing Group
Number analyzed (Participants) | 22 | 19
ridge width change (mm) | -1.41 (2.11) | -0.66 (1.55)

3. Secondary Outcome: Change in Buccal Ridge Height
Description: Ridge height measured at time of tooth extraction and grafting and again at time of implant placement. Changes in ridge height are determined (negative number signifies loss of ridge height)
Time Frame: at time of implant placement at 8-10 or 18-20 weeks following tooth extraction and grafting
Measure: Mean (Standard Deviation); unit: change in bone height (mm)
Arm/Group | 8-10 Week Healing Group | 18-20 Week Healing Group
Number analyzed (Participants) | 22 | 19
change in bone height (mm) | -1.82 (2.23) | -1.18 (1.31)

ADVERSE EVENTS:
Arm/Group | 8-10 Week Healing Group | 18-20 Week Healing Group
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 1/22 | 0/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8-10 Week Healing Group (N=22) | 18-20 Week Healing Group (N=21)
poor healing of extraction site (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No